CLINICAL TRIAL: NCT04002024
Title: A Randomized Controlled Trial of Efficiency of Moisturizer Containing Licochalcone A, Decanediol, L-carnitine and Salicylic Acid in Reducing Relapsing of Acne in Thai Acne Subjects
Brief Title: Moisturizer Containing Licochalcone A, Decanediol, L-carnitine and Salicylic Acid in Reducing Relapsing of Acne
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Beiersdorf (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Eucerine proacne
Record Dates: First submitted 2019-02-27; First posted 2019-06-28 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Acne Vulgaris; Acne
Keywords: acne vulgaris; acne; licochalcone A; decanediol; L-carnitine; salicylic acid
MeSH Terms: conditions — Acne Vulgaris | interventions — Carnitine; Salicylic Acid

STUDY DESIGN:
Intervention Model Description: Split face study. Half face is ramdomly applied moisturizer containing the active ingredients of licochalcone A, decanediol, L-carnitine, and salicylic acid. Another half face is assigned to use placebo which is moisturizer without those active ingredients.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo and Treatment Arm A (Active Comparator): The patients in treatment arm A group will be received moisturizer containing the active ingredients of licochalcone A, decanediol, L-carnitine, and salicylic acid on the right side of their face and placebo which is moisturizer without those active ingredients on the left side of their face.
  Interventions: Other: Moisturizer with active ingredients; Other: Placebo
- Treatment and Placebo Arm B (Active Comparator): The patients in treatment arm B group will be received moisturizer containing the active ingredients of licochalcone A, decanediol, L-carnitine, and salicylic acid on the left side of their face and placebo which is moisturizer without those active ingredients on the right side of their face.
  Interventions: Other: Moisturizer with active ingredients; Other: Placebo

INTERVENTIONS:
Other: Moisturizer with active ingredients — Moisturizer with active ingredients: 1 fingertip unit to cover one side of the face twice a day
  Other Names: Moisturizer containing Licochalcone A, Decanediol, L-carnitine and Salicylic Acid
Other: Placebo — Placebo: 1 fingertip unit to cover one side of the face twice a day
  Other Names: Moisturizer without those active ingredients

SUMMARY:
Moisturizer containing the active ingredients of licochalcone A, decanediol, L-carnitine, and salicylic acid may be beneficial in alternative treatment of acne in maintenance phase. This study aims to evaluate the efficacy and safety of moisturizer containing the active ingredients of licochalcone A, decanediol, L-carnitine, and salicylic acid during the maintenance phase of acne in Thai patients.

DETAILED DESCRIPTION:
Acne is a chronic inflammatory skin condition. The four main mechanisms that lead to acne include excessive production of sebum from hair follicles, sebum retention, proliferation of Propionibacterium acne, and finally inflammation. Many topical agents are available for treating acute phase of acne. However, only few such as adapalene have been proved to be beneficial in maintenance phase. New active ingredients such as licochalcone, decanediol, L-carnitine, and salicylic acid have been mentioned recently, but there are only few published studies aiming on those ingredients. This study aims to evaluate the efficacy and safety of moisturizer containing the active ingredients of licochalcone A, decanediol, L-carnitine, and salicylic acid during the maintenance phase of acne in Thai patients. This study will be divided into 2 phases: induction and maintenance phase.

Induction phase

One hundred and ten acne vulgaris patients who have mild to moderate severity according to IGA (Investigator's Global Assessment) scale for Acne Vulgaris will be treated with Epiduo® (fixed combination of adapalene 0.1%/benzoyl peroxide 2.5% gel) for 8 weeks. In moderate acne vulgaris cases, 1-2 capsules of oral doxycycline per day will be prescribed. Only patients who have at least 50 percent reduction in numbers of acne vulgaris or at least 2 grade improvement according to IGA grade from baseline will be included in maintenance phase.

Maintenance phase

Fifty patients will be treated with moisturizer containing active ingredientss on one side of the face and placebo which is moisturizer without active ingredients on the other side according to the randomization for 12 weeks. Patients will be followed up every 4 weeks (week4, week8, week12). The outcome will be assessed by

1. Acne lesion count and severity according to IGA scale.
2. Bioengineering evaluation

   * Stratum corneum hydration will be evaluated by Corneometer®
   * Transepidermal water loss will be evaluated by Tewameter®
   * Sebum will be evaluated by Sebumeter®
3. The assessment of skin dyspigmentation and skin radiance assessed by Visia® and Antera 3D®.
4. The skin tolerability (erythema, dryness, scaling, stinging/burning and pruritus)
5. Rating of satisfaction evaluted by VAS score.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who had age more than 18 years
2. Female patients must use any reliable contraceptive methods except contraceptive pills for at least 1 month prior to the study and 6 months after the completion of the study
3. Being diagnosed acne vulgaris by dermatologist. Patients will be clinically diagnosed with acne vulgaris by dermatologists by presenting of noninflammatory open or closed comedones (blackheads and whiteheads) or inflammatory lesions, which may be papules, pustules, or nodules. Lesions are likely to occur in high concentration of sebaceous glands, for example, face, neck, chest, and back.

Inclusion criteria of induction phase

1. Patients who have mild to moderate severity of acne vulgaris according to IGA* (Investigator's Global Assessment) scale of FDA (Food and Drug Administration) at both cheek and diagnosed by dermatologists.

IGA* Scale for Acne Vulgaris 0= Clear skin with no inflammatory or noninflammatory lesions

1. rare non-inflammatory lesions with no more than one small inflammatory lesion
2. mild severity defines as some non-inflammatory lesions with no more than a few inflammatory lesions (papules/ pustules only, no nodular lesions)
3. moderate severity defines as up to many non-inflammatory lesions and may have some inflammatory lesions, but no more than one small nodular lesion
4. moderate severity defines as up to many non-inflammatory lesions and may have some inflammatory lesions, but no more than one small nodular lesion
5. Severe severity defines as up to many non-inflammatory and inflammatory lesions, but no more than a few nodular lesions

Maintenance phase

1. Patients who have at least 50 percent reduction in numbers of acne vulgaris or at least 2 grade improvement according to IGA Grade from baseline

Exclusion Criteria:

1. Patients receive antibiotics, systemic treatment for acne such as isotretinoin or contraceptive pills, or spironolactone within 4 weeks prior to the study
2. Patients with active skin disease at face within 2 weeks prior to the study
3. Patients with an allergic to licochalcone A, decanediol, L-carnitine, or salicylic acid
4. Patients with severe and uncontrollable comorbidities
5. Pregnant or breastfeeding women
6. Patients with other types of acne apart from acne vulgaris
7. Patients with an allergic to oral doxycycline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Reduction of acne lesion count of moisturizer containing the active ingredients of licochalcone A, decanediol, L-carnitine, and salicylic acid | 12th week
  Acne lesion count was evaluated by counting papules, pustules and total number of inflammatory lesions between two sides of face.
Relapse rate of acne of moisturizer containing the active ingredients of licochalcone A, decanediol, L-carnitine, and salicylic acid | 12th week
  Relapse rate is defined as a percentage of patient who had acne lesion count worse more than 50%.
Time to acne relapse of moisturizer containing the active ingredients of licochalcone A, decanediol, L-carnitine, and salicylic acid | 12th week
  Time to relapse is defined as time to which patient had acne lesion count worse more than 50%.

SECONDARY OUTCOMES:
Side effects of moisturizer containing the active ingredients of licochalcone A, decanediol, L-carnitine, and salicylic acid | 12th week
  Side effects are defined as erythema, dryness, scaling, stinging, burning and pruritus.
Patients' satisfaction of moisturizer containing the active ingredients of licochalcone A, decanediol, L-carnitine, and salicylic acid | 12th week
  Satisfaction is evaluated by overall VAS score.
Efficacy of moisturizer containing the active ingredients of licochalcone A, decanediol, L-carnitine, and salicylic acid in reducing skin dyspigmentation | 12th week
  Skin dyspigmentation is evaluated by Visia® and Antera® which determined melanin and hemoglobin parameters.
Stratum corneum hydration during the use of moisturizer containing the active ingredients of licochalcone A, decanediol, L-carnitine, and salicylic acid | 12th week
  Stratum corneum hydration will be assessed by Corneometer®. The unit is Corneometer® units from 0-130.
Transepidermal water loss during the use of moisturizer containing the active ingredients of licochalcone A, decanediol, L-carnitine, and salicylic acid | 12th week
  Transepidermal water loss will be assessed by Tewameter® which reported in g/h/m2.
Skin sebum content during the use of moisturizer containingthe active ingredients of licochalcone A, decanediol, L-carnitine, and salicylic acid | 12th week
  Skin sebum content will be assessed by Sebumeter®. The unit is Sebumeter® units from 0-350 (approximated to μg/cm2 in a certain range).

CONTACTS AND LOCATIONS:
Overall Officials: Kanokvalai Kulthanan, M.D., Principal Investigator — Mahidol University
Locations (1):
- Department of Dermatology, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkoknoi, Bangkok, Thailand

REFERENCES:
- [Background] Clark AK, Saric S, Sivamani RK. Acne Scars: How Do We Grade Them? Am J Clin Dermatol. 2018 Apr;19(2):139-144. doi: 10.1007/s40257-017-0321-x. PMID 28891036
- [Background] Tan JK, Tang J, Fung K, Gupta AK, Thomas DR, Sapra S, Lynde C, Poulin Y, Gulliver W, Sebaldt RJ. Development and validation of a comprehensive acne severity scale. J Cutan Med Surg. 2007 Nov-Dec;11(6):211-6. doi: 10.2310/7750.2007.00037. PMID 18042334
- [Background] Zhang JZ, Li LF, Tu YT, Zheng J. A successful maintenance approach in inflammatory acne with adapalene gel 0.1% after an initial treatment in combination with clindamycin topical solution 1% or after monotherapy with clindamycin topical solution 1%. J Dermatolog Treat. 2004 Dec;15(6):372-8. doi: 10.1080/09546630410021702. PMID 15764049
- [Background] Thiboutot DM, Shalita AR, Yamauchi PS, Dawson C, Kerrouche N, Arsonnaud S, Kang S. Adapalene gel, 0.1%, as maintenance therapy for acne vulgaris: a randomized, controlled, investigator-blind follow-up of a recent combination study. Arch Dermatol. 2006 May;142(5):597-602. doi: 10.1001/archderm.142.5.597. PMID 16702497
- [Background] Thielitz A, Sidou F, Gollnick H. Control of microcomedone formation throughout a maintenance treatment with adapalene gel, 0.1%. J Eur Acad Dermatol Venereol. 2007 Jul;21(6):747-53. doi: 10.1111/j.1468-3083.2007.02190.x. PMID 17567301
- [Background] Dreno B, Bissonnette R, Gagne-Henley A, Barankin B, Lynde C, Kerrouche N, Tan J. Prevention and Reduction of Atrophic Acne Scars with Adapalene 0.3%/Benzoyl Peroxide 2.5% Gel in Subjects with Moderate or Severe Facial Acne: Results of a 6-Month Randomized, Vehicle-Controlled Trial Using Intra-Individual Comparison. Am J Clin Dermatol. 2018 Apr;19(2):275-286. doi: 10.1007/s40257-018-0352-y. PMID 29549588
- [Background] Bhatia N, Bhatt V, Martin G, Pillai R. Two Randomized, Double-Blind, Split-Face Studies to Compare the Irritation Potential of Two Topical Acne Fixed Combinations Over a 21-Day Treatment Period. J Drugs Dermatol. 2016 Jun 1;15(6):721-6. PMID 27272079
- [Background] Chularojanamontri L, Tuchinda P, Kulthanan K, Varothai S, Winayanuwattikun W. A double-blinded, randomized, vehicle-controlled study to access skin tolerability and efficacy of an anti-inflammatory moisturizer in treatment of acne with 0.1% adapalene gel. J Dermatolog Treat. 2016;27(2):140-5. doi: 10.3109/09546634.2015.1079298. Epub 2015 Sep 2. PMID 26293170
- [Background] Chen X, Wang S, Yang M, Li L. Chemical peels for acne vulgaris: a systematic review of randomised controlled trials. BMJ Open. 2018 Apr 28;8(4):e019607. doi: 10.1136/bmjopen-2017-019607. PMID 29705755
- [Background] Matsunaga K, Leow YH, Chan R, Kerrouche N, Paliargues F. Adjunctive usage of a non-comedogenic moisturizer with adapalene gel 0.1% improves local tolerance: a randomized, investigator-blinded, split-face study in healthy Asian subjects. J Dermatolog Treat. 2013 Aug;24(4):278-82. doi: 10.3109/09546634.2012.661037. Epub 2012 Mar 4. PMID 22384983
- [Derived] Kulthanan K, Trakanwittayarak S, Tuchinda P, Chularojanamontri L, Limphoka P, Varothai S. A Double-Blinded, Randomized, Vehicle-Controlled Study of the Efficacy of Moisturizer Containing Licochalcone A, Decanediol, L-Carnitine, and Salicylic Acid for Prevention of Acne Relapse in Asian Population. Biomed Res Int. 2020 Oct 16;2020:2857812. doi: 10.1155/2020/2857812. eCollection 2020. PMID 33150170